CLINICAL TRIAL: NCT06716593
Title: Trajectory of Body Composition Identifies Locally Advanced Gastric Cancer with Cachexia Following Neoadjuvant Chemotherapy (FJMUGS-2411)
Brief Title: Trajectory of Body Composition Identifies LAGC with Cachexia Following NACT
Acronym: FJMUGS-2411
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., M.D. FACS, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: FJMUGS-2411
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Gastric Cancer; Trajectory
Keywords: locally advanced gastric cancer; neoadjuvant chemotherapy; cachexia; CT; adjuvant chemotherapy
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This longitudinal, multicentre cohort study included LAGC patients treated with NACT between 01/2010-12/2021. BC measurements including skeletal muscle mass (SMM) and total adipose tissue area (TATA) were evaluated by computed tomography at the third lumbar vertebra at baseline and follow-up imaging. Unsupervised latent class growth mixed models were applied to distinguish potential longitudinal SMM and TATA trajectories for identifying cachexia. The primary study endpoint was overall survival (OS), with secondary endpoints including Recurrence-free survival (RFS), objective response rate (ORR) and safety. Multiple Cox proportional hazards models were used to calculate adjusted hazard ratios (HRs) for survival.

DETAILED DESCRIPTION:
This is a retrospective, longitudinal, multicenter, real-world cohort study

ELIGIBILITY:
Inclusion Criteria:(1) locally advanced gastric cancer (cT2-4NxM0) with clinical staging before neoadjuvant chemotherapy, (2) no history of other malignant tumors, (3) no evidence of distant metastasis or invasion of adjacent organs, and (4) patients who underwent radical gastrectomy following neoadjuvant chemotherapy.

-

Exclusion Criteria: (1) history of gastric surgery; (2) acute cardiovascular disease (such as cerebrovascular or coronary artery injury) within the past three months; (3) emergency surgery; (4) active infection or severe systemic immunodeficiency; and (5) incomplete serological, computed tomography, or anthropometric data.

-

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data were collected from 600 consecutive patients diagnosed with locally advanced gastric cancer (cT2-4NanyM0) between 2010, and 2021, identified at 5 tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
3-year overall survival; 5-year overall survival | 3 years or 36 months; 5 years or 60months
  Survival status at 3/5 years: survival, death, survival with tumor, deletion.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, M.D. FACS, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China